CLINICAL TRIAL: NCT05952765
Title: Evaluation of Pink Esthetic Score and Soft Tissue Changes Following Immediate Implants Using Partially Demineralized Dentin Matrix as Jumping Gap Filling Material Versus Xenograft. A Randomized Clinical Trial.
Brief Title: Pink Esthetic Score Around Immediate Implants Using PDDM as Jumping Gap Filling Material.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mihad Ibrahim, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7691
Record Dates: First submitted 2023-07-08; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Prostheses; Endosseous Dental Implant Failure
Keywords: alveolar bone; immediate implant; soft tissue changes
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The two groups will be equally prepared for both surgical procedures. Then the decision of which group will receive (PDDM), and which will receive xenograft will be taken according to the randomized numbers placed in opaque sealed envelopes. The number will be picked by the supervisor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partially demineralized dentin matrix graft (Experimental): * A high-speed fine finishing stone and saline irrigation will be used to clean extracted teeth from periodontal ligaments, soft tissue attachments, caries, and restorations if present.
  * Teeth particles will be partially demineralized using nitric acid 2% for fifteen minutes.
  * Finally, the prepared partially demineralized dentin matrix graft granules will be washed twice with distilled water and phosphate buffered saline
  * Immediate implant of appropriate dimensions will be placed and the previously prepared partially demineralized dentin matrix graft will be used to graft the jumping gap.
  * Customized healing abutment will be used.
  * In Osseo integrated implants temporary abutment will be removed and impressions for final restoration will be performed after 3 months.
  Interventions: Procedure: Immediate implant
- xenograft (Active Comparator): * After tooth extraction, thorough curettage will be performed.
  * Immediate implant of appropriate dimensions will be placed, and the jumping gap will be grafted with xenograft "Cerabone" .
  * Customized healing abutment will be used.
  * In Osseo integrated implants temporary abutment will be removed and impressions for final restoration will be performed after 3 months.
  Interventions: Procedure: Immediate implant

INTERVENTIONS:
Procedure: Immediate implant — * Local anesthesia Septanest special® will be administered prior to the procedure.
  * Teeth extraction will be initiated by intrasulcular incision via 15 C blade without flap elevation.
  * The tooth to be extracted will be luxated atraumatically using periotomes and thin straight elevator and delivered using forceps.
  * The socket will be inspected for integrity, using a UNC graduated periodontal probe.
  grafting material either experimental or control will be used to graft jumping gap.

SUMMARY:
Will there be a difference in Pink Esthetic score and soft tissue changes around immediate implants in maxillary esthetic zone following grafting the jumping gap with partially demineralized dentin matrix compared with xenograft?

DETAILED DESCRIPTION:
This study aims to evaluate the soft tissue changes as well as hard tissue changes around immediate implants in maxillary esthetic zone following grafting the jumping gap with partially demineralized dentin matrix in comparison to xenograft.

Because xenogeneic bone is so readily available in substantial quantities, it has been the subject of notable research. However, because they contain organic material from a foreign species, xenogeneic bones are inherently very antigenic.

According to experimental results, PDDM encourages bone regeneration in a manner like autogenous bone. Both cortical bone and autogenous tooth grafts share similar physical and chemical characteristics, including optimal biodegradability, not requiring a separate surgery to harvest the graft and space maintenance capabilities. PDDM is a valuable comparator to autogenous bone in ARP and around dental implants in guided bone regeneration procedures

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age; with non-restorable teeth requiring replacement with immediate implants in the maxillary esthetic zone.
* Absence of active infection at the surgical site.
* Adequate primary stability following immediate implant placement.
* Intact socket walls following the extraction.
* Class I dental socket based on a preoperative CBCT scan
* Buccal plate thickness more than 1 mm and thick biotype.
* Compliant patients who will sign an informed consent and agree to the follow up period.

Exclusion criteria

* Poor oral hygiene or the lack of regular maintenance.
* Individuals with compromised immune system or debilitating systemic disease.
* The presence of parafunctional habits (bruxism or clenching).
* External root resorption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pink esthetic score | twelve months after final restoration
  a fourteen point scale to evaluate pink esthetics. The pink esthetic score (PES) estimates the esthetic results of soft tissue surrounding the implant with regarding 7 points : mesial, distal papilla, soft tissue margin, soft tissue contour, alveolar process, colour, texture. the score of zero will be lowest and two will be the highest for each of the seven points with zero being the lowest and 14 being the highest.

SECONDARY OUTCOMES:
Vertical and horizontal radiographic changes in bone dimensions | immediate post operative and twelve months after final restoration
  cone beam CT will be used to detect vertical and horizontal changes
Midfacial mucosal alteration | preoperative and twelve months after final restoration
  rubber base impressions taken before the surgical procedure and 12 months after implant restoration. Then, casts were poured with type IV die stone and optically scanned. The obtained models were compared by digital superimposition in a matching software to measure the vertical alterations of the buccal peri-implant soft tissue.
Patient satisfaction | one year after final restoration
  a twelve point questionnaire to evaluate patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny Mostafa, Professor, Principal Investigator — Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
baseline data and follow up measurements will be shared while keeping patients' identity protected.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: till publication
Access Criteria: public